CLINICAL TRIAL: NCT06967688
Title: The Effect of Wearable Technology-Enhanced Intervention on Family Caregivers' Self-Efficacy and Quality of Life in Dementia Care
Brief Title: The Effect of Wearable Technology-Enhanced Intervention on Family Caregivers
Acronym: dementia care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Ecem Ozgul, Research Assistant, Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 223S049; 223S049 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2025-05-03; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-12

CONDITIONS: Dementia
Keywords: dementia; caregivers; telehealth; wearable technology
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartwatch-Supported Intervention (Experimental): This arm included informal caregivers of people with dementia who participated in a smartwatch-supported intervention. The intervention began with a structured interview session based on the section "Caring for Yourself as a Caregiver" from the book Caring for People with Dementia: Brief Practical Care Tips for Every Caregiver. During the initial session (lasting no more than 45 minutes), caregivers were introduced to the use of smartwatches and their various health-tracking parameters (e.g., heart rate monitoring, inactivity alerts, women's health tracking, weight tracking, blood oxygen levels, stress monitoring, water intake tracking, sleep monitoring). Caregivers were assisted in pairing the smartwatches with their smartphones and were provided with smartwatch diaries to record their health parameters and, optionally, to express their caregiving-related thoughts and feelings. Following the first meeting, weekly phone calls were conducted with each caregiver over an eight-week peri
  Interventions: Other: Smartwatch-Supported Caregiver Intervention
- Usual Care (No Intervention): This group included informal caregivers of people with dementia who did not receive any additional intervention beyond their usual caregiving routine. They continued their caregiving responsibilities as usual, without the support of wearable technologies or structured training.

INTERVENTIONS:
Other: Smartwatch-Supported Caregiver Intervention — This intervention involved informal caregivers of people with dementia using smartwatches to monitor and manage their own health parameters over an 8-week period. The primary goal was to enhance caregivers' self-efficacy and overall well-being by providing real-time health data through wearable technology. Caregivers were introduced to the smartwatch features, which included heart rate monitoring, inactivity alerts, sleep tracking, stress level monitoring, weight tracking, water intake reminders, and blood oxygen level measurements. Caregivers were instructed to track these parameters using the smartwatch and record their health behaviors in provided diaries.Weekly phone consultations lasting no more than 5 minutes were conducted throughout the 8-week intervention, where caregivers' use of the smartwatch and diaries was reviewed, and general discussions about their health and caregiving experiences took place. The intervention aimed to integrate health self-monitoring into the caregi
  Arms: Smartwatch-Supported Intervention

SUMMARY:
This study aimed to evaluate the effect of a smartwatch-supported intervention on the self-efficacy and quality of life of informal caregivers providing care to individuals with dementia. Informal caregiving, especially in dementia, poses significant psychological and physical challenges. Low self-efficacy among caregivers can negatively impact their coping skills, health behaviors, and overall quality of life. The intervention used commercially available smartwatches that provided real-time data on physical activity, sleep, and stress levels. These devices were used as part of a 8-week caregiver support program aimed at promoting better self efficacay and quality of life level of caregiver of dementia.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of a smartwatch-supported intervention on the self-efficacy and quality of life of informal caregivers providing care to individuals with dementia. Informal caregiving, especially in dementia, poses significant psychological and physical challenges. Low self-efficacy among caregivers can negatively impact their coping skills, health behaviors, and overall quality of life. The intervention used commercially available smartwatches that provided real-time data on physical activity, sleep, and stress levels. These devices were used as part of a 8-week caregiver support program aimed at promoting self-care, stress awareness, and time management. This randomized controlled trial involved 44 participants, who were assigned to either the intervention group (smartwatch-supported care) or the control group (usual care). Outcome measures included caregiver self-efficacy and quality of life, assessed both before and after the intervention using validated instruments. The study hypothesized that caregivers in the intervention group would demonstrate improved self-efficacy and better quality of life compared to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* a) Able to speak and understand Turkish, b) Primarily responsible for the care of the PwD, c) Provides at least 4 hours of care per day, d) Owns a smartphone (for smartwatch integration), e) Able to use both a mobile phone and a smartwatch (adherence tested through a descriptive characteristic form), f) Willing to participate.

Exclusion Criteria:

* a)Hospitalization of patient or caregiver due to acute condition, b) Caregiver's visual or hearing impairment, c) New diagnosis affecting caregiver's mental health (e.g., depression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
The Revised Scale for Caregiving Self-Efficacy | 0, 2, and 6 months (measured at baseline, 2 months, and 6 months)
  According to Bandura's 'Social Cognitive Learning Theory' self-efficacy refers to an individual's confidence in their ability to perform a challenging activity. This concept plays a crucial role in managing daily tasks and effectively coping with difficulties. Individuals with high self-efficacy are more motivated and resilient in facing challenges.
Short Form 36 Quality of Life Scale | 0, 2, and 6 months (measured at baseline, 2 months, and 6 months)
  Quality of life was assessed to understand the impact of the intervention on the caregivers' overall well-being. The caregivers' quality of life was measured using a validated scale that evaluated physical health, psychological well-being, social relationships, and environmental factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Balçova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, we do not plan to share individual participant data (IPD) with other researchers. The data will be kept confidential and only used for the purposes of this study.